CLINICAL TRIAL: NCT04702451
Title: Tailored vs. Anatomical Ablation Strategy for Persistent Atrial Fibrillation
Acronym: Tailored-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Volta Medical (Industry)
Collaborators: Fortrea (Industry); CardiaBase (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLIPL-01-002
Record Dates: First submitted 2021-01-07; First posted 2021-01-08 (Estimated); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation
Keywords: Persistent Atrial Fibrillation; Catheter Ablation; Electrogram dispersion
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Tailored (Experimental): Tailored ablation strategy
  Interventions: Procedure: Dispersion ablation + PVI; Device: VX1
- Anatomical (Active Comparator): Anatomical ablation strategy
  Interventions: Procedure: PVI

INTERVENTIONS:
Procedure: Dispersion ablation + PVI — Ablation of spatio-temporal dispersion electrograms in combination with pulmonary vein antrum isolation
  Arms: Tailored
Device: VX1 — VX1-based dispersion mapping
  Arms: Tailored
Procedure: PVI — Pulmonary vein antrum isolation
  Arms: Anatomical

SUMMARY:
Atrial Fibrillation (AF) ablation is typically performed in predefined anatomic regions of the left atrium without attempting to identify patient-specific areas of interest. This procedure is referred to as Pulmonary Vein Isolation (PVI).

The hypothesis in this Study is that a tailored ablation strategy targeting areas of spatio-temporal dispersion in combination with PVI is superior to an anatomical ablation strategy targeting PVI alone for the treatment of persistent AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older candidates for a first AF ablation
* Symptomatic AF, refractory to at least one antiarrhythmic medication
* Persistent or long-standing persistent AF with documentation of (ECG, Holter, physician's letter): AF duration of ≥ 3 months and ≤ 5 years (≥ 3 months and < 1 year in the United States) or 1 effective cardioversion followed by AF recurrence lasting ≥ 3 months
* Continuous anticoagulation with warfarin (INR 2-3) or NOAC for > 4 weeks prior to ablation
* Patients must be able and willing to provide written informed consent to participate in the clinical trial
* At least 60% of patients (224 patients) in persistent AF ≥ 6 months including at least 15% (56 patients) of long-standing persistent AF ≥ 12 months

Exclusion Criteria:

* Paroxysmal and short-standing AF < 3 months
* Long-standing persistent AF > 5 years (≥ 1 year in the United States)
* ≥ 2 previous ineffective cardioversion sessions in case of undetermined AF duration
* Severe obesity (BMI > 40)
* Very dilated Left Atrium (LA)(e.g. LA diameter > 60 mm and/or LA surface > 40 cm2 determined by 2D echocardiography)
* Patients with AF secondary to an obvious reversible cause
* Inadequate anticoagulation as defined in the inclusion criteria
* LA thrombus on Transesophageal Echocardiography (TEE) or CT Scan prior to procedure
* Contraindications to anticoagulation (heparin, warfarin or NOAC)
* Patients who are or may potentially be pregnant
* Previous surgical or catheter ablation for AF
* Any cardiac surgery within the past 2 months (60 days) (includes PCI)
* Myocardial infarction within the past 2 months (60 days)
* Previous atrioventricular valve surgery
* History of blood clotting or bleeding abnormalities
* Documented arterial thromboembolic event (including TIA) within the past 12 months (365 days)
* Rheumatic Heart Disease
* Chronic severe Heart Failure (NYHA functional class IV and/or LVEF < 25%)
* Awaiting cardiac transplantation or other cardiac surgery within the next 12 months (365 days)
* Unstable angina within the past month
* Acute illness or active systemic infection or sepsis
* AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause
* Diagnosed atrial myxoma
* Significant severe pulmonary disease, (e.g. patients with restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease in GOLD stage IV) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms (e.g. unstable or untreated sleep apnea)
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment
* Enrollment in an investigational study evaluating another device, biologic, or drug
* Presence of intramural thrombus, tumor or other abnormality or condition that precludes vascular access, or manipulation of the catheter
* Life expectancy or other disease processes likely to limit survival to less than 12 months
* Acute Covid-19 infection (fever and/or biological inflammatory syndrome, and positive test documented)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Deisenhofer, MD, Study Chair — Deutsches Herzzentrum Muenchen
Locations (26):
- United States (8):
  - Grandview Medical Center, Birmingham, Alabama
  - Ascension St. Vincent's, Jacksonville, Florida
  - Washington University, St Louis, Missouri
  - Northwell Health, New York, New York
  - New York Presbyterian Queens Hospital, Queens, New York
  - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Inova Fairfax, Falls Church, Virginia
- Belgium (2):
  - OLV Aalst, Aalst
  - UZ Leuven, Leuven
- France (11):
  - Pôle Santé République, Clermont-Ferrand
  - Hôpital Saint Philibert, Lomme
  - Hôpital Louis Pradel - Hospices Civils de Lyon, Lyon
  - Hôpital Saint-Joseph, Marseille
  - Hôpital Privé Jacques Cartier, Massy
  - Hôpital Privé du Confluent, Nantes
  - Clinique Saint George, Nice
  - Centre Cardiologique du Nord, Saint-Denis
  - Clinique Rhéna, Strasbourg
  - Clinique Pasteur, Toulouse
  - CHRU Nancy, Vandœuvre-lès-Nancy
- Germany (3):
  - Klinikum Coburg, Coburg
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Deutsches Herzzentrum München, München
- Netherlands (2):
  - OLVG Amsterdam, Amsterdam
  - Isala Hartcentrum Zwolle, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seitz J, Bars C, Theodore G, Beurtheret S, Lellouche N, Bremondy M, Ferracci A, Faure J, Penaranda G, Yamazaki M, Avula UM, Curel L, Siame S, Berenfeld O, Pisapia A, Kalifa J. AF Ablation Guided by Spatiotemporal Electrogram Dispersion Without Pulmonary Vein Isolation: A Wholly Patient-Tailored Approach. J Am Coll Cardiol. 2017 Jan 24;69(3):303-321. doi: 10.1016/j.jacc.2016.10.065. PMID 28104073
- [Background] Seitz J, Durdez TM, Albenque JP, Pisapia A, Gitenay E, Durand C, Monteau J, Moubarak G, Theodore G, Lepillier A, Zhao A, Bremondy M, Maluski A, Cauchemez B, Combes S, Guyomar Y, Heuls S, Thomas O, Penaranda G, Siame S, Appetiti A, Milpied P, Bars C, Kalifa J. Artificial intelligence software standardizes electrogram-based ablation outcome for persistent atrial fibrillation. J Cardiovasc Electrophysiol. 2022 Nov;33(11):2250-2260. doi: 10.1111/jce.15657. Epub 2022 Sep 18. PMID 35989543
- [Result] Deisenhofer I, Albenque JP, Busch S, Gitenay E, Mountantonakis SE, Roux A, Horvilleur J, Bakouboula B, Oza S, Abbey S, Theodore G, Lepillier A, Guyomar Y, Bessiere F, Jan Smit J, Mohr Durdez T, Milpied P, Appetiti A, Guerrero D, De Potter T, De Chillou C, Goldbarg S, Verma A, Hummel JD; TAILORED-AF Investigators. Artificial intelligence for individualized treatment of persistent atrial fibrillation: a randomized controlled trial. Nat Med. 2025 Apr;31(4):1286-1293. doi: 10.1038/s41591-025-03517-w. Epub 2025 Feb 14. PMID 39953289
- [Derived] Deisenhofer I, Seitz J, Nguyen-Tu MS, Lotteau S, Bars C, Albenque JP, Busch S, Gitenay E, Mountantonakis S, Roux A, Horvilleur J, Bakouboula B, Oza S, Abbey S, Theodore G, Lepillier A, Guyomar Y, Bessiere F, Smit JJ, Rajendra A, Cooper DH, Rashid H, De Potter T, De Chillou C, Goldbarg S, Verma A, Morales G, Milpied P, Hummel JD, Kalifa J. Women with persistent atrial fibrillation need more than pulmonary vein isolation: personalised extra-pulmonary vein ablation strategy vs. pulmonary vein isolation alone in the TAILORED-AF trial. Europace. 2025 Oct 31;27(11):euaf281. doi: 10.1093/europace/euaf281. PMID 41311304

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Among the 377 patients enrolled, 3 patients did not receive any ablation, because their ablation was cancelled or postponed. They were therefore not randomized and exited the study.
Groups:
- Tailored: Tailored ablation strategy
  Dispersion ablation + PVI: Ablation of VX1-based spatio-temporal dispersion electrograms in combination with pulmonary vein antrum isolation
Period: Overall Study
Arm/Group | Tailored | Anatomical
Started | 188 | 186
Completed | 174 | 174
Not Completed | 14 | 12

BASELINE CHARACTERISTICS:
Population: The baseline safety population included all randomized participants who underwent their first ablation procedure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailored | Anatomical | Total
Number analyzed (Participants) | 187 | 183 | 370
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (8.5) | 64.9 (8.5) | 65.7 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 35 | 77
  Male | 145 | 148 | 293
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 3 | 2 | 5
  Belgium | 6 | 4 | 10
  United States | 29 | 30 | 59
  France | 128 | 124 | 252
  Germany | 21 | 23 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Free From Documented AF After One Ablation Procedure
Description: Freedom from documented AF episodes > 30 seconds, with or without anti-arrhythmic drugs (AADs), 12 months after a single index ablation procedure
Time Frame: 12 months
Population: mITT: all randomized participants except for those who were deemed ineligible after randomization and before the ablation procedure, those who did not have any ablation procedure, and those lost to follow-up during the 3-month blanking period.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored | Anatomical
Number analyzed (Participants) | 180 | 177
Participants | 158 | 124

2. Secondary Outcome: Number of Participants Free From Documented AF/AT After One or Two Ablation Procedures
Description: Freedom from documented AF/AT episodes > 30 seconds, after one or two procedures, with or without AADs, at 12 months
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored | Anatomical
Number analyzed (Participants) | 180 | 177
Participants | 136 | 126

3. Secondary Outcome: Number of Participants Free From Documented AF/AT After One Ablation Procedure
Description: Freedom from documented AF/AT episodes > 30 seconds, with or without AADs, 12 months after a single ablation procedure
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored | Anatomical
Number analyzed (Participants) | 180 | 177
Participants | 108 | 106

4. Secondary Outcome: Number of Participants With Complications (Safety Composite Endpoint)
Description: Complications at 12 months: death, cerebrovascular events, or serious treatment-related adverse event
Time Frame: 12 months
Population: The safety population included all randomized participants who underwent their first ablation procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored | Anatomical
Number analyzed (Participants) | 187 | 183
Participants | 8 | 5

ADVERSE EVENTS:
Time Frame: 1 year after the study index ablation procedure
Arm/Group | Tailored | Anatomical
All-Cause Mortality (participants affected / at risk) | 2/187 | 0/183
Serious Adverse Events (participants affected / at risk) | 21/187 | 11/183
Other Adverse Events (participants affected / at risk) | 12/187 | 10/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tailored (N=187) | Anatomical (N=183)
Cardiac tamponade or perforation (Cardiac disorders) | 2 (2) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Severe cardiac decompensation (Cardiac disorders) | 1 (1) | 1 (1)
Puncture-site hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Transient phrenic nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fluid overload (Cardiac disorders) | 9 (9) | 3 (3)
Pericarditis or pericardial effusion (Cardiac disorders) | 4 (4) | 0 (0)
Vascular access complications (Vascular disorders) | 3 (3) | 3 (3)
Post-ablation fever (Infections and infestations) | 1 (1) | 0 (0)
Abnormal ECG requiring hospitalization (Cardiac disorders) | 0 (0) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tailored (N=187) | Anatomical (N=183)
Covid-19 (Infections and infestations) | 12 (12) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT04702451/Prot_002.pdf
  • Statistical Analysis Plan (2024-02-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT04702451/SAP_003.pdf